CLINICAL TRIAL: NCT00414102
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Demonstrate the Subjective Treatment Effects of Ramelteon on Sleep Using a Post Sleep Questionnaire - Interactive Voice Response System (PSQ-IVRS) in an "At-Home Setting" in an Adult Population With Chronic Insomnia
Brief Title: Subjective Efficacy of Ramelteon on Sleep in Adults With Chronic Insomnia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-069; U1111-1115-2043 (Registry Identifier: WHO)
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Insomnia
Keywords: Chronic Insomnia; Sleep Initiation and Maintenance Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 8mg, tablets, orally, once nightly for up to 28 days.
  Other Names: TAK-375; Rozerem™
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once nightly for up to 28 days.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the subjective treatment effects of ramelteon, once daily (QD), on sleep using a post sleep questionnaire-interactive voice response system in adults with chronic insomnia.

DETAILED DESCRIPTION:
Approximately 60 to 70 million adults in the United States alone are affected by insomnia. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating, and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia-related conditions that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism, and greater rates of accidents.

Ramelteon is marketed for the treatment of insomnia characterized by difficulty with sleep onset under the brand name of Rozerem™.

This study will be comprised of two groups of subjects, 1) an outpatient group and 2) an inpatient group. The inpatient group will be used as reference arm as previously conducted studies in the sleep laboratory setting. Study participation is anticipated to be about 50 days (approximately 1.75 months).

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Body mass index between 18 and 34, inclusive.
* Based on sleep history, has had chronic insomnia for at least 3 months.
* Based on sleep history, reports a history of subjective sleep latency greater than or equal to 60 min and a subjective total sleep time of less than or equal to 6.5 hours.
* The difference of the average subjective sleep latency from days 1-3 to days 5-7 has to be less than or equal to 20 minutes during the single blind run-in period.
* On at least 3 of the first 5 nights of single-blind run-in placebo treatment, the subject must have an subjective sleep latency of greater than or equal to 45 minutes and subjective total sleep time of less than or equal to 6.5 hours.
* Based on sleep history, habitual bedtime is between 10:00 PM and 1:00 AM.
* Willing to have a fixed bedtime and agrees to go to bed within 30 minutes of the habitual bedtime during the entire study.
* Consistent access to a touch-tone phone and are willing to complete all paper and telephone questionnaires within 60 minutes of awakening each morning throughout the entire duration of the study.
* Willing to remain in bed for at least 6.5 hours each night during the entire study.
* Based on sleep history, uses pharmacological assistance to sleep 0 to 4 times per week in the last 3 months.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin, and melatonin related compounds.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first dose of single-blind study medication, whichever is longer.
* Has sleep schedule changes required by employment (eg, shift worker) within three months prior to the administration of single-blind study medication.
* Has flown across greater than 3 time zones within 7 days prior to screening, or will travel across 2 or more time zones during the course of the study.
* Has participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the first night of single-blind study medication.
* Has ever had a history of seizures; sleep apnea, restless leg syndrome, periodic leg movement syndrome, chronic obstructive pulmonary disease, fibromyalgia, or a positive test result for the aforementioned ailments on the screening polysomnography.
* History of psychiatric disorder within the past 6 months.
* History of drug addiction or drug abuse within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised, or regularly consumes more than 14 alcoholic drinks per week, or for the inpatient subject consumed any alcoholic drinks within 24 hours of any polysomnography visits.
* Current significant hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, neurological, or metabolic disease, unless currently controlled and stable with protocol-allowed medication, within 30 days prior to the first night of single-blind study medication.
* Uses tobacco products or any other products during nightly awakenings that may interfere with the sleep wake cycle.
* Positive urine drug screen at initial screening Visit 2.
* For inpatient subjects: has a positive breathalyzer test on any of the PSG assessment visits.
* Exhibit a placebo response during single blinded placebo run in period.
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * indicate that continuation in the study would not be in the best interests of the subject.
* Positive hepatitis panel including hepatitis A virus- Immunoglobulin M, hepatitis-B surface antigen, hepatitis C virus antibody.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including the following:

  * Anxiolytics Antipsychotics
  * over-the-counter and Prescription Sedatives
  * Hypnotics
  * Narcotic analgesics
  * Antidepressants
  * Beta-blockers
  * Anticonvulsants
  * St. John's wort
  * Sedating H1 antihistamines
  * Kava-kava
  * Systemic steroids
  * Ginkgo-biloba
  * Respiratory stimulants
  * over-the-counter and prescription diet aids
  * Sedating Decongestants
  * Muscle relaxants
  * Melatonin and all other drugs or supplements known to affect sleep/wake function.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 552 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Average subjective Sleep Latency from Day 15 to Day 21 | Day 22

SECONDARY OUTCOMES:
Subjective Measures of Sleep Latency. | Weeks 1 and 2 or Final Visit
Subjective Total Sleep Time. | Weeks 1, 2 and 3 or Final Visit
Wake Time after Sleep Onset | Weeks 1, 2 and 3 or Final Visit
Number of Awakenings. | Weeks 1, 2 and 3 or Final Visit
Quality of Sleep. | Weeks 1, 2 and 3 or Final Visit
Rebound insomnia assessed from Nights 22 to 28 via self-reported sleep latency. | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research & Development Center
Locations (52):
- United States (52):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Los Angeles Area, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Denver Area, Colorado
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Kansas City Area, Kansas
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Auburn, Maine
  - Baltimore Area, Maryland
  - Washington D.C. Area, Maryland
  - Hattiesburg, Mississippi
  - Saint Louis Area, Missouri
  - Albuquerque, New Mexico
  - Long Island City, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Gallipolis, Ohio
  - Oklahoma City, Oklahoma
  - Portland Area, Oregon
  - Clarkes Summitt, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Anderson, South Carolina
  - Charleston Area, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle Area, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI